CLINICAL TRIAL: NCT06350357
Title: Conventional Clipping Versus Punching Closure for Defect Closure After ESD：a Randomized Controlled Trial
Brief Title: Conventional Clipping Versus Punching Closure
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ningbo No. 1 Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2024B014
Record Dates: First submitted 2024-04-01; First posted 2024-04-05 (Actual); Last update posted 2024-04-05 (Actual); Status verified 2024-04

CONDITIONS: the Rate of Complete Closure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- punching closure (Experimental): punching closure for defect closure after ESD
  Interventions: Other: punching closure
- Conventional clipping (Active Comparator): Conventional clipping for defect closure after ESD
  Interventions: Other: Conventional clipping

INTERVENTIONS:
Other: punching closure — The hole clamping and the grooves hold the metal clips better
  Arms: punching closure
Other: Conventional clipping — Metal lip closure is one of the most commonly used closure methods
  Arms: Conventional clipping

SUMMARY:
Endoscopic submucosal dissection (ESD) is an important minimally invasive treatment method for early digestive tract tumors, with a high cure rate, and it is widely used in clinical practice. And wound closure after ESD is a great challenge, which is closely related to postoperative perforation bleeding. Clip closure is one of the most commonly used closure methods. However, when the wound is large or when the wound is located more difficult to operate, conventional closure may lead to delayed perforation, and postoperative clips may be prone to early spontaneous shedding. The authors have recently reported a method that may be able to close larger and difficult wounds because the grooves can better fix the metal clips. The latest study suggests that this approach may be safe and effective, but the study has a small sample size and has no controls. Therefore, high-quality clinical study evidence related to punch closure is required in the strategy of defect closure after ESD, in order to better evaluate the feasibility and safety of this new endoscopic closure method.

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients undergoing gastrointestinal ESD wound closure in the First Affiliated Hospital of Ningbo University from April 20, 2024 to December 31, 2025; 2. Age 18-75 years old; 3. Patients who voluntarily agreed to participate in this study and signed informed consent.

Exclusion Criteria:

* 1. Persons under the age of 18 2. Unwilling or unable to provide informed consent 3. Treatment or radiotherapy for malignant diseases, severe chronic heart or lung diseases, coronary or cerebrovascular events requiring hospitalization within the last 3 months 4.. Severe abdominal pain, bloating, nausea and other abdominal symptoms 5.. Patients with lifelong anticoagulant therapy or severe bleeding disorders, and patients who have recently taken anticoagulant or antiplatelet drugs 6. Pregnant or lactating 7. Patients with aggressive lesions and recurrent or residual tumors

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Completely closed | 4 weeks
  The wound is completely closed without dehiscence

SECONDARY OUTCOMES:
delayed hemorrhage | 2 weeks and 4 weeks
  Any symptoms of gastrointestinal bleeding (e. g. hematochezia) occurred within 30 days after polypectomy and were classified as mild or severe according on the severity of the bleeding

CONTACTS AND LOCATIONS:
Locations (1):
- Ningbo first hospital, Ningbo, Zhejiang, China